CLINICAL TRIAL: NCT04648345
Title: Efficacy and Safety of Erector Spinal Plane Block (ESPB) for Intraoperative and Postoperative Analgesia in Laparoscopic Cholecystectomy : A Randomized, Single-blind，Controlled Clinical Trial.
Brief Title: Efficacy and Safety of Erector Spinal Plane Block (ESPB) for Analgesia in Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20004-0-01
Record Dates: First submitted 2020-11-03; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Analgesia
Keywords: erector spinal plane block; analgesia; laparoscopic cholecystectomy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: A randomized, single-blinded, controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector spinal plane block group (ESPB group) (Experimental): After induction of general anesthesia, pre-operative ultrasound-guided bilateral erector spinae plane block will be performed in the ESPB group.
  Interventions: Procedure: Erector spinal plane block
- Vertebral side block group (VSB group) (Active Comparator): After induction of general anesthesia, pre-operative ultrasound-guided bilateral vertebral side block will be performed in the VSB group.
  Interventions: Procedure: Erector spinal plane block
- Local block group （LB group） (Placebo Comparator): Local block will be performed at the surgical incisions after the surgery under general anesthesia.
  Interventions: Procedure: Erector spinal plane block

INTERVENTIONS:
Procedure: Erector spinal plane block — After induction of general anesthesia, pre-operative ultrasound-guided bilateral erector spinae plane block/ vertebral side block will be performed in the ESPB/VSB group. Local block will be performed at the surgical incisions after the surgery under general anesthesia. All the intervention will be performed without patients' awareness.
  Other Names: Vertebral side block; Local block

SUMMARY:
Purpose: to evaluate the efficacy and safety of erector spinal block (ESB) for analgesia in laparoscopic cholecystectomy（LC）.

Method: This study is a randomized, single-blind, controlled clinical trial. Pre-operative ultrasound-guided bilateral erector spinae plane block will be performed in the ESPB group. Vertebral side block will be performed in the VSB group. And the control group will receive local anaesthesia after the surgery. Intraoperative and postoperative analgesia effect and side effects will be compared between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1-3
* Scheduled for elective laparoscopic cholecystectomy surgery under general anesthesia

Exclusion Criteria:

* patient refusal
* pregnancy
* history of allergy to study drugs
* neurological and cognitive disorders
* coagulopathy
* chronic pain disorders
* infections at the injection site
* history of abdominal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Pain intensity at rest(Hour 2) | Hour 2
  Using the Numeric Rating Scale (NRS) to evaluate the pain intensity at rest two hours after the surgery.
Pain intensity at rest (Hour 6) | Hour 6
  Using the Numeric Rating Scale (NRS) to evaluate the pain intensity at rest six hours after the surgery.
Pain intensity at rest (Hour 24) | Hour 24
  Using the Numeric Rating Scale (NRS) to evaluate the pain intensity at rest 24 hours after the surgery.

SECONDARY OUTCOMES:
The overall dose of remifentanil | During the surgery
  The overall dose of remifentanil used in the surgery.

IPD SHARING:
Plan to Share IPD: No